CLINICAL TRIAL: NCT02058368
Title: A Randomized, Double-blind, Parallel Group Study to Compare the Efficacy and Safety of Combination Treatment With Dutasteride (0.5mg) and Tamsulosin (0.2mg) With Tamsulosin (0.2mg) Monotherapy, Administered Once Daily for 2 Years, on the Improvement of Symptoms and Health Outcomes in Men With Moderate to Severe Benign Prostatic Hyperplasia
Brief Title: Study to Compare the Efficacy and Safety of Combination Treatment With Dutasteride and Tamsulosin With Tamsulosin Monotherapy, in Men With Moderate to Severe Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114265
Record Dates: First submitted 2014-01-23; First posted 2014-02-10 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Quality of Life
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Run-in phase: All subjects qualifying for the study will entered into a placebo run-in phase will receive one soft gelatin placebo capsule (swallowed whole and not chewed) and one oral disintegrating placebo tablet once daily (OD) (dissolved on the tongue then swallowed not chewed), following the first meal each day for four weeks. Randomized treatment phase: Subjects will be instructed to take 1 dutasteride 0.5 milligram (mg) capsule (swallowed whole and not chewed) and one tamsulosin 0.2mg tablet OD (dissolved on the tongue then swallowed not chewed) following the first meal each day for 104 weeks.
  Interventions: Drug: Dutasteride 0.5mg capsules; Drug: Dutasteride placebo capsules; Drug: Tamsulosin 0.2mg tablets; Drug: Disintegrating placebo tamsulosin tablet
- Arm 2 (Experimental): Run-in phase: All subjects qualifying for the study will entered into a placebo run-in phase will receive one soft gelatine placebo capsule (swallowed whole and not chewed) and one oral disintegrating placebo tablet OD (dissolved on the tongue then swallowed not chewed), following the first meal each day for four weeks. Randomized treatment phase: Subjects will be instructed to take 1 placebo dutasteride 0.5mg capsule (swallowed whole and not chewed) and one tamsulosin 0.2mg tablet OD (dissolved on the tongue then swallowed not chewed) following the first meal each day for 104 weeks.
  Interventions: Drug: Dutasteride placebo capsules; Drug: Tamsulosin 0.2mg tablets; Drug: Disintegrating placebo tamsulosin tablet

INTERVENTIONS:
Drug: Dutasteride 0.5mg capsules — Dutasteride 0.5mg capsules will be supplied as plain, oblong, opaque, dull yellow soft gelatin capsules.
  Arms: Arm 1
Drug: Dutasteride placebo capsules — Dutasteride placebo will be supplied as plain, oblong, opaque, dull yellow soft gelatin capsules.
Drug: Tamsulosin 0.2mg tablets — Commercially available tamsulosin 0.2mg tablets will be supplied.
Drug: Disintegrating placebo tamsulosin tablet — Disintegrating placebo tamsulosin tablet will be supplied for the run-in period.

SUMMARY:
This is a multicentre, randomised, double-blind, parallel group study in Asian subjects. The aim of the study is to investigate whether combination therapy with dutasteride and tamsulosin is more effective than tamsulosin monotherapy for the improvement of symptoms and health outcomes in an at risk population of benign prostatic hyperplasia (BPH) clinical progression including older men (>=50 years), with moderate-severe symptoms of BPH, enlarged prostates (>=30 cubicentimeter [cc]) and prostate specific antigen (PSA) >= 1.5 nanograms per milliliter (ng/mL). Each subject who met the eligibility criteria at screening will enter a four-week single-blind, placebo run-in period following which each subject will be randomised into a 2 year double-blind treatment phase. The total study duration for each subject will be up to 110 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged >=50 years
* Clinical diagnosis of BPH by medical history and physical examination, including a digital rectal examination (DRE)
* International Prostate Symptom Score (IPSS) >=12 points at Screening
* Prostate volume >=30cc (by TRUS)
* Total serum Prostate Specific Antigen (PSA) >=1.5ng/mL and <= 10 ng/mL at Screening
* Maximum urinary flow rate (Qmax) >5mL/sec and 15mL/sec and minimum voided volume of >=125 milliliter (mL) at Screening
* Asparate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Fluent and literate in local language with the ability to comprehend and record information on the IPSS, BPH-related Health Status (BHS), BPH Impact Index (BII), and Problem Assessment Scale Sexual Function Inventory (PAS- SFI) questionnaires
* Men with a female partner of childbearing potential must agree to use a condom up to 6 months after the last dose (applies only to countries where the local product monograph for dutasteride mandates condom use for men with a female partner of childbearing potential)

Exclusion Criteria:

* History or evidence of prostate cancer (e.g. positive biopsy or ultrasound, suspicious Digital Rectal Examination [DRE]). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable PSA are eligible for the study. Note: If total serum PSA is >4ng/mL and unless PSA value has been stable for at least the past 2 years, the investigator should make every appropriate effort to exclude the possibility of prostate cancer, including consideration of prostate biopsy.
* Previous prostatic surgery (including TURP, laser, transrectal high intensity focused ultrasounds(HIFU), thermotherapy, transurethral needle ablation (TUNA), balloon dilatation, and stent replacement) or other invasive procedures to treat BPH.
* History of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days prior to the Screening Visit. Catheterisation (<10F) is acceptable with no time restriction.
* History of AUR within 3 months prior to Screening Visit.
* Post-void residual volume >250mL (suprapubic ultrasound) at Screening.
* Any conditions other than BPH, which may in the judgment of the investigator, result in urinary symptoms or changes in flow rate (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, or acute or chronic urinary tract infections).
* Unstable liver disease (chronic stable hepatitis B and C are acceptable if subject meets entry criteria).
* History of renal insufficiency, or serum creatinine >1.5 times the upper limit of normal at Screening.
* Any unstable, serious co-existing medical condition(s) including, but not limited to:

  1. Myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
  2. Postural hypotension, dizziness, vertigo or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
  3. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to study procedures in the opinion of the investigator or GSK medical monitor. Investigator may consult with GSK Medical Monitor if condition could interfere with subject's safety
  4. History of breast cancer or clinical breast examination finding suggestive of malignancy.
  5. History of malignancy within the past five years, except for basal cell carcinoma of the skin. Subjects with a priori malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Current or Previous Use of the following medications:

  1. Use of any 5-alpha-reductase inhibitor (e.g. finasteride), any drugs with antiandrogenic properties (e.g. spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, progestational agents), or other drugs noted for gynaecomastia effects, or that could affect prostate volume, within the 6 months preceding the historical TRUS or Screening Visit and throughout the study (other than as study medication). Previous use of dutasteride should not be within 6 months of the baseline or historical TRUS.
  2. Anabolic steroids (subject must discontinue for 6 months prior to study entry to be eligible) and agree not to take them for the duration of the study.
  3. Phytotherapy for BPH within 2 weeks of Screening Visit and/or predicted to need phytotherapy during the study.
  4. Use of any alpha-adrenoreceptor blockers within 2 weeks of Screening Visit (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin, doxazosin, silodosin) and/or predicted to need any alpha blockers other than the study prescribed tamsulosin.
  5. Use of any alpha-adrenoreceptor agonists (e.g. pseudoephedrine, phenylephedrine, ephedrine) or anticholinergics (e.g. oxybutynin,tolterodine, darifenacin, solifenacin,propantheline) or cholinergics (e.g. bethanecol chloride) within 48 hours prior to all uroflowmetry assessments.
* Hypersensitivity to any alpha-/beta- adrenoreceptor blocker or 5-alpha-reductase inhibitor, or other chemically-related drugs.
* Participation in any investigational or marketed drug trial within 30 days (or 5 half-lives of drug, whichever is the longer) preceding the Screening Visit and/or plans to participate in such a trial during the course of this study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- China (9):
  - GSK Investigational Site, Xiame, Fujian
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
- Japan (8):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamanashi
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
- Taiwan (7):
  - GSK Investigational Site, Chiayi City
  - GSK Investigational Site, Hualien City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Kaohsiung Hsien
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Tau-Yuan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Haque N, Masumori N, Sakamoto S, Ye Z, Yoon SJ, Kuo HC, Brotherton B, Wilson T, Muganurmath C, McLaughlin M, Manyak M. Superiority of dutasteride 0.5 mg and tamsulosin 0.2 mg for the treatment of moderate-to-severe benign prostatic hyperplasia in Asian men. Int J Urol. 2018 Nov;25(11):944-951. doi: 10.1111/iju.13785. Epub 2018 Sep 9. PMID 30198102
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, parallel group trial to assess the effectiveness and safety of dutasteride (Dut) 0.5 milligram (mg) and tamsulosin (Tam) 0.2 mg combination compared to Tam 0.2 mg. The study consisted of a single-blind, placebo run-in, followed by a 2 year treatment. Eligible subjects were randomized to Dut + Tam or Dut placebo + Tam
Pre-assignment Details: Six hundred and fifty moderate to severe benign prostatic hyperplasia (BPH) subjects were screened with 607 participants receiving as least one dose of the study medication (China 243, Japan 135, Korea 181, Taiwan 48). Five hundred and twelve subjects completed the study with 95 subjects withdrawn.
Groups:
- Placebo +Tam 0.2mg: Participants were randomized in a ratio of 1:1 to receive Dut placebo QD plus Tam 0.2 mg QD for 104 Weeks.
- Dut 0.5 mg + Tam 0.2 mg: Participants were randomized in a ratio of 1:1 to receive Dut 0.5 mg QD plus Tam 0.2 mg QD for 104 Weeks.
Period: Overall Study
Arm/Group | Placebo +Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Started | 302 | 305
Completed | 261 | 251
Not Completed | 41 | 54
Not completed — Adverse Event | 15 | 20
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 0 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 22 | 26

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population, comprised of all randomized participants who received or did not receive study treatment
Groups:
- Placebo + Tam 0.2mg: Participants were randomized in a ratio of 1:1 to receive Dut placebo QD plus Tam 0.2 mg QD for 104 Weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg | Total
Number analyzed (Participants) | 302 | 305 | 607
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Intent-to-Treat Population, comprised of all randomized participants who received or did not receive study treatment
  Years | 66.2 (6.85) | 66.8 (6.82) | 66.5 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent-to-Treat Population, comprised of all randomized participants who received or did not receive study treatment
  Participants
    Female | 0 | 0 | 0
    Male | 302 | 305 | 607
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent-to-Treat Population, comprised of all randomized participants who received or did not receive study treatment
  Participants
    Asian - East Asian Heritage | 234 | 236 | 470
    Asian - Japanese Heritage | 68 | 67 | 135
    Asian - Southeast Asian Heritage | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) by Last Observation Carried Forward (LOCF) Approach at 24 Months
Description: IPSS (also called IPSS total score) is the sum of the seven questions with each score ranging from 0 (best) to 5 (worst). IPSS was self administered at screening, Baseline and each time-point of Month 3, 6, 9, 12, 15, 18, 21 and 24. Seven questions included are incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. The total IPSS score can range from 0-35 with severity catagories of mild (0 to 7), moderate (8 to 19) or severe (20 to 35). LOCF is defined as carrying forward the last non-missing post-Baseline assessment for participants with missing visit data and/or for participants who discontinued from the study. Baseline value is defined as the latest non-missing assessment of either treatment start date or randomization date. Month 24 is the primary timepoint and earlier timepoints are considered secondary. Change from Baseline defined as difference between Post-Baseline value and Baseline value.
Time Frame: Baseline and 3, 6, 9, 12, 15, 18, 21 and 24 months
Population: ITT Population.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Score on scale
  Month 3, n=299, 296: number analyzed (Participants) | 299 | 296
  Month 3, n=299, 296 | -4.07 (0.34) | -3.28 (0.34)
  Month 6, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 6, n=300, 298 | -3.73 (0.37) | -3.36 (0.37)
  Month 9, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9, n=300, 298 | -4.14 (0.36) | -4.28 (0.36)
  Month 12,n= 300, 298: number analyzed (Participants) | 300 | 298
  Month 12,n= 300, 298 | -3.93 (0.36) | -4.30 (0.36)
  Month 15, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15, n=300, 298 | -3.95 (0.36) | -4.90 (0.36)
  Month 18, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18, n=300, 298 | -3.84 (0.38) | -4.54 (0.38)
  Month 21, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21, n=300, 298 | -3.94 (0.38) | -4.66 (0.38)
  Month 24, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24, n=300, 298 | -3.53 (0.39) | -4.96 (0.39)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.069, General linear model — Change from Baseline = Treatment + Country + Baseline Value. P-values for Dut 0.5 mg + Tam 0.2 mg versus Placebo + Tam 0.2mg are based on t-tests from the general linear model. Reported means are model based adjusted means; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.06 to 1.65] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 3
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.43, General linear model — Change from Baseline = Treatment + Country + Baseline Value. P-values for Dut 0.5 mg + Tam 0.2 mg versus Placebo + Tam 0.2 mg are based on t-tests from the general linear model. Reported means are model based adjusted means; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.55 to 1.29] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 6
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.76, General linear model — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.05 to 0.77] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 9
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.41, General linear model — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.27 to 0.53] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 12
Statistical Analysis 5: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.039, General linear model — Change from Baseline = Treatment + Country + Baseline Value. P-values for Dut 0.5 mg+Tam 0.2 mg versus Placebo+ Tam 0.2 mg are based on t-tests from the general linear model. Reported means are model based adjusted means; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.85 to -0.05] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 15
Statistical Analysis 6: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.15, General linear model — [p-value comment as in outcome 1, analysis 5]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.65 to 0.26] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 18
Statistical Analysis 7: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.15, General linear model — [p-value comment as in outcome 1, analysis 5]; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.68 to 0.25] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 21
Statistical Analysis 8: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.004, General linear model — [p-value comment as in outcome 1, analysis 5]; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-2.40 to -0.46] — Estimates are based on adjusted means from the general linear model. The adjusted mean difference was based on combination minus tamsulosin monotherapy for Month 24

2. Secondary Outcome: Percent Change in Prostate Volume From Baseline
Description: Prostate Volume measurements were conducted annually using Transrectal ultrasound (TRUS). The following calculation was utilized to assess the prostate volume (cc): pi/6 (Anteroposterior Width multiplied by Cephalocaudal Width multiplied by Transverse Width). Post-Baseline prostate volume was calculated at 12 and 24 months. Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline was reported based on the LOCF. Change from Baseline defined as difference between Post-Baseline value and Baseline value and reported as a percentage.
Time Frame: Baseline,12 and 24 months
Population: ITT Population.
Measure: Mean (Standard Error); unit: Cubic centimeters (cc)
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Cubic centimeters (cc)
  Month 12, n=287, 286: number analyzed (Participants) | 287 | 286
  Month 12, n=287, 286 | 0.2 (1.28) | -22.8 (0.99)
  Month 24, n=287, 286: number analyzed (Participants) | 287 | 286
  Month 24, n=287, 286 | 3.6 (1.45) | -24.8 (1.06)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Log(Post-Baseline Prostate Volume / Baseline Prostate Volume) = Log(Baseline Prostate Volume) + Treatment + Country. P-values are based on t-tests from the general linear model; Mean Difference (Final Values) = -23.0, 95% CI 2-sided [-25.9 to -20.1], Standard Error of Mean 1.48 — The adjusted mean estimates, adjusted mean differences, and confidence intervals are expressed in terms of percentage change from Baseline for Month 12
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority — Estimates are based on the adjusted means from the general linear model: Log(Post-Baseline Prostate Volume / Baseline Prostate Volume) = Log(Baseline Prostate Volume) + Treatment + Country. P-values are based on t-tests from the general linear model; p < .001, General linear model; Mean Difference (Final Values) = -28.4, 95% CI 2-sided [-31.7 to -25.2], Standard Error of Mean 1.65 — The adjusted mean estimates, adjusted mean differences, and confidence intervals are expressed in terms of percentage change from Baseline for Month 24

3. Secondary Outcome: Number of Participants With IPSS Improvement From Baseline
Description: Improvement in IPSS was categorized as improvement, no change and worsening. Improvement defined as greater than or equal to 2 points, greater than or equal to 3 points and greater than or equal to 25 percent in participants at months 3,6,9,12,15,18,21 and 24 . Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline was reported based on the LOCF. Change from Baseline defined as difference between Post-Baseline value and Baseline value.
Time Frame: Baseline and 3, 6, 9,12,15,18,21 and 24 months
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Month 3,>= 3 units, n=299, 296: number analyzed (Participants) | 299 | 296
  Month 3,>= 3 units, n=299, 296 | 160 | 157
  Month 3,>= 2 units, n=299,296: number analyzed (Participants) | 299 | 296
  Month 3,>= 2 units, n=299,296 | 190 | 176
  Month 3,>= 25percent, n=299, 296: number analyzed (Participants) | 299 | 296
  Month 3,>= 25percent, n=299, 296 | 134 | 123
  Month 6,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 6,>= 3 units, n=300, 298 | 156 | 156
  Month 6,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 6,>= 2 units, n=300, 298 | 179 | 176
  Month 6,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 6,>= 25percent, n=300, 298 | 131 | 133
  Month 9,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9,>= 3 units, n=300, 298 | 157 | 177
  Month 9,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9,>= 2 units, n=300, 298 | 185 | 193
  Month 9,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9,>= 25percent, n=300, 298 | 128 | 150
  Month 12,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 12,>= 3 units, n=300, 298 | 154 | 171
  Month 12,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 12,>= 2 units, n=300, 298 | 179 | 191
  Month 12,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 12,>= 25percent, n=300, 298 | 131 | 154
  Month 15,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15,>= 3 units, n=300, 298 | 171 | 186
  Month 15,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15,>= 2 units, n=300, 298 | 186 | 203
  Month 15,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15,>= 25percent, n=300, 298 | 133 | 160
  Month 18,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18,>= 3 units, n=300, 298 | 156 | 171
  Month 18,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18,>= 2 units, n=300, 298 | 173 | 187
  Month 18,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18,>= 25percent, n=300, 298 | 136 | 148
  Month 21,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21,>= 3 units, n=300, 298 | 169 | 178
  Month 21,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21,>= 2 units, n=300, 298 | 186 | 194
  Month 21,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21,>= 25percent, n=300, 298 | 141 | 161
  Month 24,>= 3 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24,>= 3 units, n=300, 298 | 156 | 184
  Month 24,>= 2 units, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24,>= 2 units, n=300, 298 | 175 | 197
  Month 24,>= 25percent, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24,>= 25percent, n=300, 298 | 137 | 169
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.91, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 3
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.31, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 3
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.42, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 3
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.92, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 6
Statistical Analysis 5: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.89, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 6
Statistical Analysis 6: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.81, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 6
Statistical Analysis 7: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.080, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 9
Statistical Analysis 8: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.42, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 9
Statistical Analysis 9: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.060, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 9
Statistical Analysis 10: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.14, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 12
Statistical Analysis 11: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.26, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 12
Statistical Analysis 12: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.048, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 12
Statistical Analysis 13: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.17, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 15
Statistical Analysis 14: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.11, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 15
Statistical Analysis 15: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.022, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 15
Statistical Analysis 16: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.18, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 18
Statistical Analysis 17: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.19, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 18
Statistical Analysis 18: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.28, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 18
Statistical Analysis 19: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.39, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 21
Statistical Analysis 20: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.42, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 21
Statistical Analysis 21: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.084, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 21
Statistical Analysis 22: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.016, Mantel Haenszel — P-value for IPSS improvement >= 3 units has been presented for Month 24
Statistical Analysis 23: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.047, Mantel Haenszel — P-value for IPSS improvement >= 2 units has been presented for Month 24
Statistical Analysis 24: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.007, Mantel Haenszel — P-value for IPSS improvement >= 25 percent has been presented for Month 24

4. Secondary Outcome: Change From Baseline in Maximum Urine Flow Rate (Qmax) by LOCF Approach
Description: Qmax is defined as maximum urine flow. Qmax was measured with Uroflow meter (Urodyn 1000) at Screening, Baseline, and at Months 6,12,18 and 24. Change from Baseline Qmax at each scheduled post-Baseline assessment was compared in terms of combination treatment (Dut plus Tam) versus tamsulosin treatment using t-tests from a general linear model with effects for treatment, country, and Baseline Qmax. Baseline value was defined as the latest non-missing assessment either treatment start date or randomization date. Change from Baseline defined as difference between Post-Baseline value and Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, 6, 12, 18 and 24 Months
Population: ITT Population
Measure: Mean (Standard Error); unit: milliliter per second (mL/sec)
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
milliliter per second (mL/sec)
  Month 6, n=270, 274: number analyzed (Participants) | 270 | 274
  Month 6, n=270, 274 | 0.62 (0.26) | 1.54 (0.26)
  Month 12, n=286, 287: number analyzed (Participants) | 286 | 287
  Month 12, n=286, 287 | 0.63 (0.28) | 1.62 (0.27)
  Month 18, n=287, 288: number analyzed (Participants) | 287 | 288
  Month 18, n=287, 288 | 0.90 (0.33) | 2.36 (0.33)
  Month 24, n=287,290: number analyzed (Participants) | 287 | 290
  Month 24, n=287,290 | 0.93 (0.32) | 2.27 (0.32)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.006, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 6; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [0.26 to 1.56], Standard Error of Mean 0.33 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.005, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 12; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [0.30 to 1.69], Standard Error of Mean 0.35 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 18; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [0.63 to 2.29], Standard Error of Mean 0.42 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 24; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [0.54 to 2.15], Standard Error of Mean 0.41 — The adjusted mean difference was based on Dut+Tam minus Tam

5. Secondary Outcome: Number of Participants With Qmax Improvement From Baseline by LOCF Approach.
Description: Qmax change from Baseline was presented using six improvement levels: >0 milliliter per second (mL/sec) and >=1 mL/sec through >=5mL/sec. Qmax percentage change from Baseline was presented using six improvement levels: >0%, >=10%, >=20%, >=30%, >=40%, and >=50%. Here, Qmax improvement of >= 3 mL/sec and Qmax percentage of >= 30 % for 24 Months has been summarized. Baseline value is defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline defined as difference between Post-Baseline value and Baseline value. Baseline value is defined as the latest non-missing assessment of either treatment start date or randomization date.
Time Frame: Baseline 6, 12, 18 and 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Month 6, >= 3 mL/sec, n=270, 274: number analyzed (Participants) | 270 | 274
  Month 6, >= 3 mL/sec, n=270, 274 | 69 | 86
  Month 6, >= 3 %, n=270, 274: number analyzed (Participants) | 270 | 274
  Month 6, >= 3 %, n=270, 274 | 70 | 86
  Month 12, >= 3 mL/sec, n=286, 287: number analyzed (Participants) | 286 | 287
  Month 12, >= 3 mL/sec, n=286, 287 | 64 | 102
  Month 12, >= 3 %, n=286, 287: number analyzed (Participants) | 286 | 287
  Month 12, >= 3 %, n=286, 287 | 73 | 107
  Month 18, >= 3 mL/sec, n=287, 288: number analyzed (Participants) | 287 | 288
  Month 18, >= 3 mL/sec, n=287, 288 | 80 | 115
  Month 18, >= 3 %, n= 287, 288: number analyzed (Participants) | 287 | 288
  Month 18, >= 3 %, n= 287, 288 | 81 | 111
  Month 24, >= 3 mL/sec, n=287, 290: number analyzed (Participants) | 287 | 290
  Month 24, >= 3 mL/sec, n=287, 290 | 77 | 121
  Month 24, >= 30 %, n=287, 290: number analyzed (Participants) | 287 | 290
  Month 24, >= 30 %, n=287, 290 | 71 | 119
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.13, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 3 mL/sec for Month 6
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.15, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 30 % for Month 6
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 3 mL/sec for Month 12
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.003, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 30 % for Month 12
Statistical Analysis 5: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.002, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 3 mL/sec for Month 18
Statistical Analysis 6: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.009, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 30 % for Month 18
Statistical Analysis 7: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 3 mL/sec for Month 24
Statistical Analysis 8: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, Mantel Haenszel — P-value for Dut+Tam vs. Tam is based on a Mantel-Haenszel test controlling for country for >= 30 % for Month 24

6. Secondary Outcome: Number of Participants With Acute Urinary Retention (AUR) or Benign Prostatic Hyperplasia (BPH)-Related Prostatic Surgery
Description: AUR is defined as condition when the participant is unable to urinate and requires bladder catheterization. AUR or BPH-related surgery event details per participant was summarized as first occurring of either AUR or BPH-related surgery.
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Overall | 15 | 4
  Year 1 subset | 8 | 2
  Year 2 subset | 7 | 2
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.012, Log Rank — Relative Risk (hazard ratio) for Dut+Tam vs. Tam is based on the Cox Proportional Hazards Model with stratification by country; Cox Proportional Hazard = 0.27, 95% CI 2-sided [0.09 to 0.81]

7. Secondary Outcome: Number of Subjects With AUR
Description: AUR is defined as condition when the participant is unable to urinate and requires bladder catheterization.
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Overall | 13 | 2
  Year 1 subset | 8 | 2
  Year 2 subset | 5 | 0
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.005, Log Rank — [p-value comment as in outcome 6, analysis 1]; Cox Proportional Hazard = 0.15, 95% CI 2-sided [0.03 to 0.68]

8. Secondary Outcome: Number of Participants With BPH-related Surgery
Description: BPH-related interventions were recorded. BPH-related interventions included adenomectomy, balloon dilatation, electroresection, thermotherapy (microwave or radiofrequency), laser resection, prostatectomy, prostatotomy, transurethral resection of the prostate, transurethral drainage of prostatic abscess, drainage of prostatic cysts, radioactive seeding of the prostate, prostatic urethral stenting, incision of periurethral stricture, ethanol injections into the prostate, transrectal high intensity focussed ultrasound, transurethral needle ablation and transurethral microwave thermotherapy.
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Overall | 3 | 2
  Year 1 subset | 0 | 0
  Year 2 subset | 3 | 2
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.68, Log Rank — [p-value comment as in outcome 6, analysis 1]; Cox Proportional Hazard = 0.69, 95% CI 2-sided [0.11 to 4.11]

9. Secondary Outcome: Change From Baseline in the BPH-related Health Status (BHS) by LOCF Approach
Description: BHS was collected as Question 8 the IPSS questionnaire regarding quality of life due to urinary symptom with scores values ranging from 0 (delightful) to 6 (terrible). Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from baseline BHS at each scheduled post-baseline assessment was compared in terms of combination treatment (Dut plus Tam) versus tamsulosin treatment using t-tests from a general linear model with effects for treatment, country, and Baseline BHS.
Time Frame: Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 Months
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Scores on scale
  Month 3, n=299, 296: number analyzed (Participants) | 299 | 296
  Month 3, n=299, 296 | -0.88 (0.08) | -0.85 (0.08)
  Month 6, n=300,298: number analyzed (Participants) | 300 | 298
  Month 6, n=300,298 | -0.89 (0.08) | -0.73 (0.08)
  Month 9, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9, n=300, 298 | -1.08 (0.08) | -0.95 (0.08)
  Month 12, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 12, n=300, 298 | -0.87 (0.08) | -0.90 (0.08)
  Month 15, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15, n=300, 298 | -0.93 (0.08) | -1.02 (0.08)
  Month 18, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18, n=300, 298 | -0.92 (0.08) | -1.00 (0.08)
  Month 21, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21, n=300, 298 | -1.08 (0.09) | -1.02 (0.09)
  Month 24, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24, n=300, 298 | -1.00 (0.08) | -1.16 (0.08)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.83, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Country + Baseline Value for Month 3; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.17 to 0.21], Standard Error of Mean 0.10 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.11, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Country + Baseline Value for Month 6; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.04 to 0.36], Standard Error of Mean 0.10 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.21, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Country + Baseline Value for Month 9; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.07 to 0.34], Standard Error of Mean 0.11 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.80, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Country + Baseline Value for Month 12; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.23 to 0.18], Standard Error of Mean 0.10 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 5: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.37, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 15; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.30 to 0.11], Standard Error of Mean 0.10 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 6: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.44, General linear model — [p-value comment as in outcome 4, analysis 3]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.30 to 0.13], Standard Error of Mean 0.11 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 7: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.60, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value for Month 21; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.16 to 0.28], Standard Error of Mean 0.11 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 8: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.16, General linear model — [p-value comment as in outcome 4, analysis 4]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.37 to 0.06], Standard Error of Mean 0.11 — The adjusted mean difference was based on Dut+Tam minus Tam

10. Secondary Outcome: Change From Baseline in BPH Impact Index (BII) by LOCF Approach
Description: The BII consists of four questions and BII total score is the sum of four questions. Total score range is 0 (no problem) to 13 (worst value). Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline BII at each scheduled post-baseline assessment was compared in terms of combination treatment (Dut plus Tam) versus tamsulosin treatment using t-tests from a general linear model with effects for treatment, country, and Baseline BII. Change from Baseline was summarized using LOCF approaches.
Time Frame: Baseline 3, 6, 9, 12, 15, 18, 21 and 24 Months
Population: ITT Population.
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Scores on scale
  Month 3, n=299, 296: number analyzed (Participants) | 299 | 296
  Month 3, n=299, 296 | -1.48 (0.14) | -1.23 (0.14)
  Month 6, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 6, n=300, 298 | -1.28 (0.15) | -1.08 (0.16)
  Month 9, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 9, n=300, 298 | -1.55 (0.15) | -1.26 (0.16)
  Month 12, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 12, n=300, 298 | -1.39 (0.16) | -1.24 (0.16)
  Month 15, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 15, n=300, 298 | -1.30 (0.16) | -1.41 (0.16)
  Month 18, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 18, n=300, 298 | -1.16 (0.16) | -1.28 (0.16)
  Month 21, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 21, n=300, 298 | -1.12 (0.17) | -1.27 (0.17)
  Month 24, n=300, 298: number analyzed (Participants) | 300 | 298
  Month 24, n=300, 298 | -1.02 (0.17) | -1.48 (0.17)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.17, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value. P-values for Dut+Tam versus Tam are based on t-tests from the general linear model; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.11 to 0.62], Standard Error of Mean 0.18 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 3
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.33, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.20 to 0.59], Standard Error of Mean 0.20 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 6
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.15, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.10 to 0.68], Standard Error of Mean 0.20 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 9
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.46, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.25 to 0.55], Standard Error of Mean 0.21 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 12
Statistical Analysis 5: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.59, General linear model — [p-value comment as in outcome 10, analysis 1]; Median Difference (Final Values) = -0.11, 95% CI 2-sided [-0.51 to 0.29], Standard Error of Mean 0.21 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 15
Statistical Analysis 6: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.56, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.52 to 0.28], Standard Error of Mean 0.20 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 18
Statistical Analysis 7: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.51, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.56 to 0.28], Standard Error of Mean 0.21 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 21
Statistical Analysis 8: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.034, General linear model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.88 to -0.03], Standard Error of Mean 0.21 — The adjusted mean difference was based on Dut+Tam minus Tam for Month 24

11. Secondary Outcome: Change From Baseline in Problem Assessment Scale of the Sexual Function Inventory (PAS-SFI)
Description: PAS SFI consists of three questions each with a range of 0 (Big Problem) to 4 (No Problem). PAS SFI was administered at screening, Baseline and at each month 12 and 24. The total PSI is the sum of the three questions; the total score range is 0 to 12. Change from Baseline PAS SFI at each scheduled post-baseline assessment was compared in terms of combination treatment (Dut plus Tam) versus tamsulosin treatment using t-tests from a general linear model with effects for treatment, country, and Baseline PAS SFI. Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline defined as difference between Post-Baseline value and Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, 12 and 24 Months
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Scores on scale
  Month 12, n=291, 293: number analyzed (Participants) | 291 | 293
  Month 12, n=291, 293 | 0.11 (0.21) | -0.91 (0.20)
  Month 24, n=291, 294: number analyzed (Participants) | 291 | 294
  Month 24, n=291, 294 | -0.11 (0.21) | -0.82 (0.21)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Country + Baseline Value.P-values for Dut+Tam versus Tam are based on t-tests from the general linear model for Month 12; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.54 to -0.50], Standard Error of Mean 0.26 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.009, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Country + Baseline Value. P-values for Dut+Tam versus Tam are based on t-tests from the general linear model for Month 24; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.23 to -0.18], Standard Error of Mean 0.27 — The adjusted mean difference was based on Dut+Tam minus Tam

12. Secondary Outcome: Number of Hospitalization Days
Description: Duration of hospitalization days due to AUR or BPH-related surgery was recorded.
Time Frame: Up to 24 Months
Population: ITT Population. Only those participants with data available at specific time point were analyzed
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 5 | 3
Days | 10.0 [6 to 18] | 9.0 [7 to 12]

13. Secondary Outcome: Number of Participants in a Hospital Ward
Description: Details of number of participants in different types of wards was recorded. Types of wards included general ward, recovery, intensive care unit, multiple ward types and others
Time Frame: Up to 24 Months
Population: ITT Population. Only those participants with data available at specific time point were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 3 | 1
Participants
  General ward | 2 | 0
  Recovery | 0 | 1
  Other | 1 | 0

14. Secondary Outcome: Number of Participants With Hospital Admissions
Description: Details of participants who were admitted to hospitals related to AUR or BPH-Related surgery has been recorded.
Time Frame: Up to 24 Months
Population: ITT Population. Only those participants with data available at specific time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 11 | 3
Participants
  Out-patient | 5 | 0
  In-patient | 6 | 3

15. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AE) and Serious AE (SAE)
Description: An adverse event is defined as any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as resulting in death, life threatening, requires hospitalization or prolongation of hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation that is medically important, All events of possible drug-induced liver injury with hyperbilirubinaemia, male breast cancer and spontaneous abortion of a female partner of a male subject
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Any Non-serious AE | 203 | 208
  Any SAE | 52 | 49

16. Secondary Outcome: Change From Baseline in Serum Prostate Specific Antigen (PSA)
Description: Total serum PSA concentrations were assessed at pre-screening, month 6, 12 and 24. Change from baseline total PSA was compared in terms of combination treatment (Dut plus Tam) versus tamsulosin treatment at each scheduled post-baseline assessment using a general linear model with effects for treatment and baseline total PSA. Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline defined as difference between Post-Baseline value and Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline 6, 12 and 24 Months
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
nanogram/milliliter (ng/mL)
  Month 6, n=292, 294: number analyzed (Participants) | 292 | 294
  Month 6, n=292, 294 | 0.2 (0.09) | -1.7 (0.08)
  Month 12, n=293, 294: number analyzed (Participants) | 293 | 294
  Month 12, n=293, 294 | 0.2 (0.08) | -1.9 (0.08)
  Month 24, n=293, 295: number analyzed (Participants) | 293 | 295
  Month 24, n=293, 295 | 0.7 (0.16) | -2.0 (0.16)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Baseline Value for Month 6; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.1 to -1.6], Standard Error of Mean 0.12 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline = Treatment + Baseline Value for Month 12; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-2.3 to -1.9], Standard Error of Mean 0.11 — The adjusted mean difference was based on Dut+Tam minus Tam
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p < .001, General linear model — Estimates are based on the adjusted means from the general linear model: Change from Baseline =Treatment + Baseline Value for Month 24; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-3.1 to -2.2], Standard Error of Mean 0.23 — The adjusted mean difference was based on Dut+Tam minus Tam

17. Secondary Outcome: Number of Participants With Vital Signs Exceeding Threshold Values
Description: Vital signs included assessment of systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate. Threshold ranges for SBP ranged from < 80 mmHg (millimeter of mercury) (lower) to > 165 mmHg (upper); for DBP ranged from < 40 mmHg (lower) to > 105 mmHg (upper) and heart rate < 40 beats per minute (bpm) (lower) to > 100 bpm (upper).
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  SBP, < 80 mmHg | 0 | 0
  SBP, > 165 mmHg | 10 | 13
  SBP, either threshold | 10 | 13
  DBP, < 40 mmHg | 0 | 0
  DBP, > 105 mmHg | 6 | 2
  DBP, either threshold | 6 | 2
  Heart rate, < 40 bpm | 0 | 0
  Heart rate, > 100 bpm | 11 | 14
  Heart rate, either threshold | 11 | 14

18. Secondary Outcome: Change From Baseline in Post Void Residual Volume
Description: Post void residual volume was measured suprapubically by ultrasound (immediately following the urinary flow measurement). Post void residual volume change from Baseline distribution at each scheduled post-Baseline assessment was compared with combination treatment (Dut plus Tam) versus tamsulosin treatment using a nonparametric van Elteren test. Baseline value was defined as the latest non-missing assessment of either treatment start date or randomization date. Change from Baseline defined as difference between Post-Baseline value and Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, 6, 12, 18 and 24 Months
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
mL
  Month 6, n=288, 290: number analyzed (Participants) | 288 | 290
  Month 6, n=288, 290 | -4.8 (52.59) | -3.0 (59.56)
  Month 12, n=291, 292: number analyzed (Participants) | 291 | 292
  Month 12, n=291, 292 | 1.5 (60.94) | -1.4 (59.19)
  Month 18, n=291, 292: number analyzed (Participants) | 291 | 292
  Month 18, n=291, 292 | -2.6 (55.67) | -1.3 (63.98)
  Month 24, n=291, 292: number analyzed (Participants) | 291 | 292
  Month 24, n=291, 292 | 2.6 (64.71) | -2.6 (62.01)
Statistical Analysis 1: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.77, Van Elteren test — P-value for Dut+Tam vs. Tam is based on a van Elteren test with stratification by country for Month 6
Statistical Analysis 2: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.84, Van Elteren test — P-value for Dut+Tam vs. Tam is based on a van Elteren test with stratification by country for Month 12
Statistical Analysis 3: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.98, Van Elteren test — P-value for Dut+Tam vs. Tam is based on a van Elteren test with stratification by country for Month 18
Statistical Analysis 4: Comparison: Placebo + Tam 0.2mg vs Dut 0.5 mg + Tam 0.2 mg; Test type: Superiority; p = 0.28, Van Elteren test — P-value for Dut+Tam vs. Tam is based on a van Elteren test with stratification by country for Month 24

19. Secondary Outcome: Number of Participants With Threshold Hematology Value.
Description: The threshold laboratory values are defined in terms of a multiplicative factor of the testing laboratory's normal range. A laboratory value that is above the upper limit factor multiplied by the upper limit of the normal (ULN) range is considered a high threshold value. A laboratory value that is below the lower limit factor multiplied by the lower limit of the normal (LLN) range is considered a low threshold value. Hematology laboratory parameters assessed included hemoglobin (Hgb), platelet count, white blood cell count (WBC) and red blood cell (RBC) count. Threshold factors are in the below table. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Hgb, <0.75 X LLN, n=287, 291: number analyzed (Participants) | 287 | 291
  Hgb, <0.75 X LLN, n=287, 291 | 0 | 0
  Platelet count, <0.75 X LLN, n=284, 283: number analyzed (Participants) | 284 | 283
  Platelet count, <0.75 X LLN, n=284, 283 | 6 | 1
  Platelet count, >1.50 X ULN, n=285, 285: number analyzed (Participants) | 285 | 285
  Platelet count, >1.50 X ULN, n=285, 285 | 0 | 0
  RBC, <0.50 X LLN, n=287, 291: number analyzed (Participants) | 287 | 291
  RBC, <0.50 X LLN, n=287, 291 | 0 | 0
  WBC, <0.50 X LLN, n=287, 291: number analyzed (Participants) | 287 | 291
  WBC, <0.50 X LLN, n=287, 291 | 0 | 0
  WBC, >3.00 X ULN, n=287, 291: number analyzed (Participants) | 287 | 291
  WBC, >3.00 X ULN, n=287, 291 | 0 | 0

20. Secondary Outcome: Number of Participants With Threshold Clinical Chemistry Value.
Description: Clinical chemistry laboratory parameters assessed included albumin, alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), creatinine, glucose, potassium, sodium, total bilirubin, total protein and urea/blood urea nitrogen (BUN). Threshold factors are in the below table. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to 24 Months
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  albumin, <0.90 X LLN, n=289, 292: number analyzed (Participants) | 289 | 292
  albumin, <0.90 X LLN, n=289, 292 | 0 | 0
  albumin, >1.20 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  albumin, >1.20 X ULN, n=289, 292 | 0 | 0
  ALT, >3.00 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  ALT, >3.00 X ULN, n=289, 292 | 0 | 0
  ALP, > 1.50 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  ALP, > 1.50 X ULN, n=289, 292 | 0 | 0
  AST, >3.00 X ULN, n=288, 292: number analyzed (Participants) | 288 | 292
  AST, >3.00 X ULN, n=288, 292 | 0 | 1
  creatinine, <0.50 X LLN, n=289, 292: number analyzed (Participants) | 289 | 292
  creatinine, <0.50 X LLN, n=289, 292 | 0 | 0
  creatinine, >3.00 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  creatinine, >3.00 X ULN, n=289, 292 | 0 | 0
  glucose, <0.70 X LLN, n=288, 292: number analyzed (Participants) | 288 | 292
  glucose, <0.70 X LLN, n=288, 292 | 0 | 0
  glucose, >1.75 X ULN, n=280, 285: number analyzed (Participants) | 280 | 285
  glucose, >1.75 X ULN, n=280, 285 | 13 | 13
  potassium, <0.75 X LLN, n=288, 292: number analyzed (Participants) | 288 | 292
  potassium, <0.75 X LLN, n=288, 292 | 0 | 0
  potassium, >1.40 X ULN, n=288, 292: number analyzed (Participants) | 288 | 292
  potassium, >1.40 X ULN, n=288, 292 | 0 | 0
  sodium, <0.90 X LLN, n=289, 292: number analyzed (Participants) | 289 | 292
  sodium, <0.90 X LLN, n=289, 292 | 0 | 0
  sodium, >1.15 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  sodium, >1.15 X ULN, n=289, 292 | 0 | 0
  total bilirubin, >2.50 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  total bilirubin, >2.50 X ULN, n=289, 292 | 0 | 0
  total protein, <0.80 X LLN, n=289, 292: number analyzed (Participants) | 289 | 292
  total protein, <0.80 X LLN, n=289, 292 | 0 | 0
  total protein, >1.15 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  total protein, >1.15 X ULN, n=289, 292 | 0 | 0
  Urea/BUN, <0.50 X LLN, n=289, 292: number analyzed (Participants) | 289 | 292
  Urea/BUN, <0.50 X LLN, n=289, 292 | 0 | 0
  Urea/BUN, >2.00 X ULN, n=289, 292: number analyzed (Participants) | 289 | 292
  Urea/BUN, >2.00 X ULN, n=289, 292 | 0 | 0

21. Secondary Outcome: Number of Participants With Digital Rectal Examination (DRE)
Description: DRE evaluation was carried out from normal/diffusely enlarged at Baseline to focal abnormalities at any time post-Baseline. DRE was assessed at screening visit, Month 6, 12, 18 , 24 and final assessment is the latest post-Baseline evaluation that was available. Here, participants with focal abnormalities are summarized. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: 6, 12, 18 , 24 months and final assessment
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Month 6, n=287, 285: number analyzed (Participants) | 287 | 285
  Month 6, n=287, 285 | 11 | 9
  Month 12, n=279, 272: number analyzed (Participants) | 279 | 272
  Month 12, n=279, 272 | 10 | 11
  Month 18, n=267, 258: number analyzed (Participants) | 267 | 258
  Month 18, n=267, 258 | 6 | 12
  Month 24, n=261, 252: number analyzed (Participants) | 261 | 252
  Month 24, n=261, 252 | 10 | 13
  Final Assessment, n=296, 295: number analyzed (Participants) | 296 | 295
  Final Assessment, n=296, 295 | 10 | 15

22. Secondary Outcome: Number of Participants With Clinically Significant Qualitative Breast Examination
Description: Qualitative breast examination included palpable breast tissue and nipple tenderness. Here, participants with clinically significant abnormalities for palpable breast tissue and nipple tenderness are summarized. Qualitative breast examination was done at screening visit, Month 6, 12, 18 , 24 and final assessment (latest post-Baseline evaluation that was available). Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: 6, 12, 18 , 24 months and final assessment
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Palpable breast tissue, Month 6, n=289, 284: number analyzed (Participants) | 289 | 284
  Palpable breast tissue, Month 6, n=289, 284 | 0 | 0
  Nipple tenderness,Month 6, n=289, 284: number analyzed (Participants) | 289 | 284
  Nipple tenderness,Month 6, n=289, 284 | 0 | 0
  Palpable breast tissue, Month 12, n=279, 273: number analyzed (Participants) | 279 | 273
  Palpable breast tissue, Month 12, n=279, 273 | 1 | 2
  Nipple tenderness,Month 12, n=279, 273: number analyzed (Participants) | 279 | 273
  Nipple tenderness,Month 12, n=279, 273 | 0 | 1
  Palpable breast tissue, Month 18, n=267, 258: number analyzed (Participants) | 267 | 258
  Palpable breast tissue, Month 18, n=267, 258 | 1 | 0
  Nipple tenderness,Month 18, n=267, 258: number analyzed (Participants) | 267 | 258
  Nipple tenderness,Month 18, n=267, 258 | 0 | 0
  Palpable breast tissue, Month 24, n=262, 252: number analyzed (Participants) | 262 | 252
  Palpable breast tissue, Month 24, n=262, 252 | 0 | 0
  Nipple tenderness, Month 24, n=262, 252: number analyzed (Participants) | 262 | 252
  Nipple tenderness, Month 24, n=262, 252 | 0 | 0
  Palpable breast tissue,final assessment, n=296,296: number analyzed (Participants) | 296 | 296
  Palpable breast tissue,final assessment, n=296,296 | 0 | 0
  Nipple tenderness,final assessment, n=296, 296: number analyzed (Participants) | 296 | 296
  Nipple tenderness,final assessment, n=296, 296 | 0 | 0

23. Secondary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior
Description: Suicidality was assessed utilizing the Columbia Suicide Severity Rating Scale (C-SSRS). It included tabular summaries of suicidal ideation and suicidal behavior questions that were administered. Assessments were carried out at Screening, Month 6, Month 12, and Month 24 (or end of treatment) visits. C-SSRS included Question1-2 were for suicidal ideation Question 1: Passive: wish to be dead, Question 2: Active: Non-specific (no method, intent or plan). Questions 6-10 were for suicidal behavior, Question 6: Preparatory Acts or Behavior, Question 7: any aborted attempt, Question 8: Any interrupted attempts, Question 9: Any non-fatal actual suicide attempt, Question 10: Completed suicide. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: 6, 12, 18 , 24 months and final assessment
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
Number analyzed (Participants) | 302 | 305
Participants
  Month 6, Suicidal ideation, Q1, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal ideation, Q1, n=289, 285 | 0 | 0
  Month 6, Suicidal ideation, Q2, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal ideation, Q2, n=289, 285 | 0 | 0
  Month 6, Suicidal behavior, Q6, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal behavior, Q6, n=289, 285 | 0 | 0
  Month 6, Suicidal behavior, Q7, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal behavior, Q7, n=289, 285 | 0 | 0
  Month 6, Suicidal behavior, Q8, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal behavior, Q8, n=289, 285 | 0 | 0
  Month 6, Suicidal behavior, Q9, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal behavior, Q9, n=289, 285 | 0 | 0
  Month 6, Suicidal behavior, Q10, n=289, 285: number analyzed (Participants) | 289 | 285
  Month 6, Suicidal behavior, Q10, n=289, 285 | 0 | 0
  Month 12, Suicidal ideation, Q1, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal ideation, Q1, n=279, 273 | 0 | 0
  Month 12, Suicidal ideation, Q2, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal ideation, Q2, n=279, 273 | 0 | 0
  Month 12, Suicidal behavior, Q6, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal behavior, Q6, n=279, 273 | 0 | 0
  Month 12, Suicidal behavior, Q7, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal behavior, Q7, n=279, 273 | 0 | 0
  Month 12, Suicidal behavior, Q8, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal behavior, Q8, n=279, 273 | 0 | 0
  Month 12, Suicidal behavior, Q9, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal behavior, Q9, n=279, 273 | 0 | 0
  Month 12, Suicidal behavior, Q10, n=279, 273: number analyzed (Participants) | 279 | 273
  Month 12, Suicidal behavior, Q10, n=279, 273 | 0 | 0
  Month 24, Suicidal ideation, Q1, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 24, Suicidal ideation, Q1, n=261, 251 | 0 | 1
  Month 24, Suicidal ideation, Q2, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 24, Suicidal ideation, Q2, n=261, 251 | 0 | 0
  Month 12, Suicidal behavior, Q6, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 12, Suicidal behavior, Q6, n=261, 251 | 0 | 0
  Month 12, Suicidal behavior, Q7, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 12, Suicidal behavior, Q7, n=261, 251 | 0 | 0
  Month 12, Suicidal behavior, Q8, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 12, Suicidal behavior, Q8, n=261, 251 | 0 | 0
  Month 12, Suicidal behavior, Q9, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 12, Suicidal behavior, Q9, n=261, 251 | 0 | 0
  Month 12, Suicidal behavior, Q10, n=261, 251: number analyzed (Participants) | 261 | 251
  Month 12, Suicidal behavior, Q10, n=261, 251 | 0 | 0
  Final assessment, Suicidal ideation,Q1, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal ideation,Q1, n=288, 285 | 0 | 1
  Final assessment, Suicidal ideation,Q2, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal ideation,Q2, n=288, 285 | 0 | 0
  Final assessment, Suicidal behavior,Q6, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal behavior,Q6, n=288, 285 | 0 | 0
  Final assessment, Suicidal behavior,Q7, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal behavior,Q7, n=288, 285 | 0 | 0
  Final assessment, Suicidal behavior,Q8, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal behavior,Q8, n=288, 285 | 0 | 0
  Final assessment, Suicidal behavior,Q9, n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal behavior,Q9, n=288, 285 | 0 | 0
  Final assessment, Suicidal behavior,Q10,n=288, 285: number analyzed (Participants) | 288 | 285
  Final assessment, Suicidal behavior,Q10,n=288, 285 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Participants who withdrew for sexual function events were followed up for 6 months after treatment discontinuation.
Arm/Group | Placebo + Tam 0.2mg | Dut 0.5 mg + Tam 0.2 mg
All-Cause Mortality (participants affected / at risk) | 1/302 | 2/305
Serious Adverse Events (participants affected / at risk) | 52/302 | 49/305
Other Adverse Events (participants affected / at risk) | 203/302 | 208/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Tam 0.2mg (N=302) | Dut 0.5 mg + Tam 0.2 mg (N=305)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 7 (7) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (3) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Ulnar nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 2 (2)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (2) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Infarction (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1)
Implant site inflammation (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Tam 0.2mg (N=302) | Dut 0.5 mg + Tam 0.2 mg (N=305)
Nasopharyngitis (Infections and infestations) | 30 (46) | 37 (45)
Upper respiratory tract infection (Infections and infestations) | 38 (72) | 24 (44)
Bronchitis (Infections and infestations) | 11 (11) | 8 (8)
Periodontitis (Infections and infestations) | 7 (9) | 6 (7)
Conjunctivitis (Infections and infestations) | 10 (10) | 2 (2)
Pharyngitis (Infections and infestations) | 10 (12) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 2 (3)
Helicobacter infection (Infections and infestations) | 2 (2) | 2 (2)
Dermatophytosis of nail (Infections and infestations) | 1 (1) | 2 (3)
Epididymitis (Infections and infestations) | 1 (1) | 2 (2)
Hordeolum (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Dacryocanaliculitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Trachoma (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Myringitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 10 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (13) | 7 (8)
Constipation (Gastrointestinal disorders) | 3 (3) | 13 (13)
Chronic gastritis (Gastrointestinal disorders) | 10 (10) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 6 (7)
Dental caries (Gastrointestinal disorders) | 8 (8) | 3 (3)
Gastritis (Gastrointestinal disorders) | 5 (6) | 5 (6)
Toothache (Gastrointestinal disorders) | 6 (7) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 2 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone formation increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus tarsi syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 16 (18) | 14 (16)
Headache (Nervous system disorders) | 10 (12) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 3 (3)
Lacunar infarction (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (3)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysmetria (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Amnestic disorder (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 7 (8)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (9) | 4 (4)
Nocturia (Renal and urinary disorders) | 2 (2) | 8 (10)
Dysuria (Renal and urinary disorders) | 6 (6) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 5 (5) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 5 (5)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 6 (7) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 2 (2)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema nummular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 7 (7)
Chest discomfort (General disorders) | 5 (5) | 5 (6)
Chest pain (General disorders) | 6 (8) | 2 (2)
Asthenia (General disorders) | 1 (2) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Gait deviation (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 8 (8) | 4 (4)
Dry eye (Eye disorders) | 4 (5) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 2 (2)
Eye discharge (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2)
Xerophthalmia (Eye disorders) | 1 (1) | 1 (1)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0)
Borderline glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Conjunctival cyst (Eye disorders) | 1 (1) | 0 (0)
Conjunctival deposit (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Lacrimation decreased (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Ciliary body disorder (Eye disorders) | 0 (0) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Iris disorder (Eye disorders) | 0 (0) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1)
Entropion (Eye disorders) | 1 (1) | 0 (0)
Corneal exfoliation (Eye disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Epicondylitis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pharyngeal injury 0 0 1 1 (<1%) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 14 (14)
Ejaculation failure (Reproductive system and breast disorders) | 1 (1) | 8 (8)
Sexual dysfunction (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Retrograde ejaculation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Organic erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Seminal vesicle atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 9 (9) | 7 (7)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 2 (2)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Microangiopathy (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral circulatory failure (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (8) | 7 (9)
Libido decreased (Psychiatric disorders) | 1 (1) | 4 (4)
Sleep disorder (Psychiatric disorders) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Disinhibition (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Tobacco abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Prostatic specific antigen increased (Investigations) | 3 (3) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1)
Lipids increased (Investigations) | 0 (0) | 1 (1)
Protein urine absent (Investigations) | 1 (1) | 0 (0)
Semen volume decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Renal scan abnormal (Investigations) | 0 (0) | 1 (1)
Residual urine volume increased (Investigations) | 0 (0) | 1 (1)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Auditory disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Late onset hypogonadism syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02058368/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02058368/SAP_001.pdf